CLINICAL TRIAL: NCT00387062
Title: Computer-Based Training in Patients With Post-Chemotherapy Cognitive Impairment, A Pilot Study
Brief Title: Computer-Based Training in Patients With Post-Chemotherapy Cognitive Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: OUT-113-2005; 06140-01
Record Dates: First submitted 2006-10-10; First posted 2006-10-12 (Estimated); Last update posted 2008-06-24 (Estimated); Status verified 2008-06

CONDITIONS: Breast Cancer; Cognitive Symptoms; Memory Disorders
Keywords: Breast Cancer; Cognitive Impairment; Chemofog; Chemobrain; Post-chemotherapy cognitive impairment
MeSH Terms: conditions — Breast Neoplasms; Neurobehavioral Manifestations; Memory Disorders; Cognitive Dysfunction; Chemotherapy-Related Cognitive Impairment

INTERVENTIONS:
Device: Computer-based Cognitive Training

SUMMARY:
The investigators hypothesize that continuous active interaction with environments that are demanding to sensory, cognitive, and motor systems, together with imbedded rewards for successful performance, will help improve memory and cognitive functioning in patients suffering from "chemobrain".

DETAILED DESCRIPTION:
Breast cancer is the most common malignancy in women in the United States, with an estimated 211,240 new cases of invasive breast cancer diagnosed among women, and 1,700 diagnosed in men, in 2005. While cure rates have improved significantly, chemotherapy for breast cancer is associated with a number of negative side effects. One of which is a deficit in cognitive function, a condition commonly referred to as "chemobrain". While the debate about cognitive decline being a result of chemotherapy is still ongoing, there is clear evidence of cognitive decline in women with breast cancer post-chemotherapy. Cognitive decline is often reported to affect memory, attention, executive functioning and information processing speed.

Studies suggest that incidence of "chemobrain" ranges from 17% - 75% in women who have undergone chemotherapy.This cognitive impairment affects quality of life by impacting patients' ability to concentrate, make decisions and to fulfill family, career, and community responsibilities.

Although there is uncertainty about the mechanisms that can lead to this cognitive decline, there is a pressing need to identify interventions that will alleviate its symptoms and help breast cancer survivors recover their cognitive functioning and resume their roles and activities at the pre-cancer level.

Brain plasticity refers to the brain's capacity for physical and functional change; it is this capacity that explains how experience induces learning throughout life. On the basis of a growing body of literature in the fields of psychophysics, neurology, neuropsychology, and brain plasticity, we hypothesize that the brain processing machinery can be refined, elaborated, and strengthened through rigorous training and learning. The purpose of this study is to investigate if such training can improve cognitive functioning.

We hypothesize that continuous active interaction with environments that are demanding to sensory, cognitive, and motor systems, together with imbedded rewards for successful performance will help improve memory and cognitive functioning in patients suffering from "chemobrain".

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older at the time of consent.
* Diagnosis of invasive breast cancer or recurrence warranting treatment with chemotherapeutic agents in the past 5 years.
* Cognitive decline, as reported by the patient, friends, or family.
* Fluent English speaker.
* Willing and able to commit to the 6-month time requirement of the entire study period.
* Willing to provide informed consent
* Willing to participate in training of the program.
* Agrees to weekly contact

Exclusion Criteria:

* Severe hearing impairments that would:

  * limit the ability to receive instructions and support; and
  * hinder performance on the computer training program.
* Self-report of untreated Axis I or II disorders (with the exception of depression, anxiety disorders, and panic disorders).
* Self-report of current diagnosis or history of major neurological illness including, but not limited to:

  * Alzheimer's disease
  * Parkinson's disease
  * Multiple sclerosis
  * Amyotrophic lateral sclerosis
* History of a stroke, transient ischemic attack (TIA) or traumatic brain injury within the past year; or lifetime history of stroke, TIA, or traumatic brain injury that has left residual expressive or receptive language problems.
* Self-report of fibromyalgia or symptoms of tremor severe enough to prevent the use of a computer mouse or other pointing device.
* Unwillingness to complete the required assessments.
* Patient is not capable of giving informed consent or unable to comprehend and/or follow instructions.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Examination of the quantitative training program progression data
Safety

SECONDARY OUTCOMES:
Quality of life health assessments
Functional outcomes assessments
Perceived stress assessments

CONTACTS AND LOCATIONS:
Overall Officials: Henry W Mahncke, PhD, Principal Investigator — Posit Science Corporation
Locations (1):
- Posit Science Corporation, San Francisco, California, United States

REFERENCES:
- [Background] Shilling V, Jenkins V. Self-reported cognitive problems in women receiving adjuvant therapy for breast cancer. Eur J Oncol Nurs. 2007 Feb;11(1):6-15. doi: 10.1016/j.ejon.2006.02.005. Epub 2006 Jul 17. PMID 16844416
- [Background] Wefel JS, Lenzi R, Theriault R, Buzdar AU, Cruickshank S, Meyers CA. 'Chemobrain' in breast carcinoma?: a prologue. Cancer. 2004 Aug 1;101(3):466-75. doi: 10.1002/cncr.20393. PMID 15274059
- [Background] Tannock IF, Ahles TA, Ganz PA, Van Dam FS. Cognitive impairment associated with chemotherapy for cancer: report of a workshop. J Clin Oncol. 2004 Jun 1;22(11):2233-9. doi: 10.1200/JCO.2004.08.094. PMID 15169812
- [Background] Schagen SB, Muller MJ, Boogerd W, Rosenbrand RM, van Rhijn D, Rodenhuis S, van Dam FS. Late effects of adjuvant chemotherapy on cognitive function: a follow-up study in breast cancer patients. Ann Oncol. 2002 Sep;13(9):1387-97. doi: 10.1093/annonc/mdf241. PMID 12196364
- [Background] van Dam FS, Schagen SB, Muller MJ, Boogerd W, vd Wall E, Droogleever Fortuyn ME, Rodenhuis S. Impairment of cognitive function in women receiving adjuvant treatment for high-risk breast cancer: high-dose versus standard-dose chemotherapy. J Natl Cancer Inst. 1998 Feb 4;90(3):210-8. doi: 10.1093/jnci/90.3.210. PMID 9462678
- [Background] Schagen SB, van Dam FS, Muller MJ, Boogerd W, Lindeboom J, Bruning PF. Cognitive deficits after postoperative adjuvant chemotherapy for breast carcinoma. Cancer. 1999 Feb 1;85(3):640-50. doi: 10.1002/(sici)1097-0142(19990201)85:33.0.co;2-g. PMID 10091737
- [Background] Brezden CB, Phillips KA, Abdolell M, Bunston T, Tannock IF. Cognitive function in breast cancer patients receiving adjuvant chemotherapy. J Clin Oncol. 2000 Jul;18(14):2695-701. doi: 10.1200/JCO.2000.18.14.2695. PMID 10894868
- [Background] Jansen CE, Miaskowski C, Dodd M, Dowling G. Chemotherapy-induced cognitive impairment in women with breast cancer: a critique of the literature. Oncol Nurs Forum. 2005 Mar 5;32(2):329-42. doi: 10.1188/05.ONF.329-342. PMID 15759070
- [Background] Paraska K, Bender CM. Cognitive dysfunction following adjuvant chemotherapy for breast cancer: two case studies. Oncol Nurs Forum. 2003 May-Jun;30(3):473-8. doi: 10.1188/03.ONF.473-478. PMID 12719746
- [Background] Wefel JS, Lenzi R, Theriault RL, Davis RN, Meyers CA. The cognitive sequelae of standard-dose adjuvant chemotherapy in women with breast carcinoma: results of a prospective, randomized, longitudinal trial. Cancer. 2004 Jun 1;100(11):2292-9. doi: 10.1002/cncr.20272. PMID 15160331
- [Background] O'Shaughnessy J. Chemotherapy-related cognitive dysfunction in breast cancer. Semin Oncol Nurs. 2003 Nov;19(4 Suppl 2):17-24. doi: 10.1053/j.soncn.2003.09.002. PMID 14702917
- [Background] Gilbert CD, Sigman M, Crist RE. The neural basis of perceptual learning. Neuron. 2001 Sep 13;31(5):681-97. doi: 10.1016/s0896-6273(01)00424-x. PMID 11567610
- [Background] Morse R, Rodgers J, Verrill M, Kendell K. Neuropsychological functioning following systemic treatment in women treated for breast cancer: a review. Eur J Cancer. 2003 Nov;39(16):2288-97. doi: 10.1016/s0959-8049(03)00600-2. PMID 14556919
- [Background] de Jong N, Candel MJ, Schouten HC, Abu-Saad HH, Courtens AM. Course of mental fatigue and motivation in breast cancer patients receiving adjuvant chemotherapy. Ann Oncol. 2005 Mar;16(3):372-82. doi: 10.1093/annonc/mdi095. Epub 2005 Jan 27. PMID 15677622
- [Background] Bender CM, Sereika SM, Berga SL, Vogel VG, Brufsky AM, Paraska KK, Ryan CM. Cognitive impairment associated with adjuvant therapy in breast cancer. Psychooncology. 2006 May;15(5):422-30. doi: 10.1002/pon.964. PMID 16097037
- [Background] Tchen N, Juffs HG, Downie FP, Yi QL, Hu H, Chemerynsky I, Clemons M, Crump M, Goss PE, Warr D, Tweedale ME, Tannock IF. Cognitive function, fatigue, and menopausal symptoms in women receiving adjuvant chemotherapy for breast cancer. J Clin Oncol. 2003 Nov 15;21(22):4175-83. doi: 10.1200/JCO.2003.01.119. PMID 14615445
- [Background] Ahles TA, Saykin A. Cognitive effects of standard-dose chemotherapy in patients with cancer. Cancer Invest. 2001;19(8):812-20. doi: 10.1081/cnv-100107743. PMID 11768035
- [Background] Bender CM, Paraska KK, Sereika SM, Ryan CM, Berga SL. Cognitive function and reproductive hormones in adjuvant therapy for breast cancer: a critical review. J Pain Symptom Manage. 2001 May;21(5):407-24. doi: 10.1016/s0885-3924(01)00268-8. PMID 11369162
- [Background] Jansen CE, Miaskowski C, Dodd M, Dowling G, Kramer J. A metaanalysis of studies of the effects of cancer chemotherapy on various domains of cognitive function. Cancer. 2005 Nov 15;104(10):2222-33. doi: 10.1002/cncr.21469. PMID 16206292
- [Background] Watters JM, Yau JC, O'Rourke K, Tomiak E, Gertler SZ. Functional status is well maintained in older women during adjuvant chemotherapy for breast cancer. Ann Oncol. 2003 Dec;14(12):1744-50. doi: 10.1093/annonc/mdg497. PMID 14630679
- [Background] Phillips KA, Bernhard J. Adjuvant breast cancer treatment and cognitive function: current knowledge and research directions. J Natl Cancer Inst. 2003 Feb 5;95(3):190-7. doi: 10.1093/jnci/95.3.190. PMID 12569140
- [Background] Cimprich B, So H, Ronis DL, Trask C. Pre-treatment factors related to cognitive functioning in women newly diagnosed with breast cancer. Psychooncology. 2005 Jan;14(1):70-8. doi: 10.1002/pon.821. PMID 15386786
- [Background] Falleti MG, Sanfilippo A, Maruff P, Weih L, Phillips KA. The nature and severity of cognitive impairment associated with adjuvant chemotherapy in women with breast cancer: a meta-analysis of the current literature. Brain Cogn. 2005 Oct;59(1):60-70. doi: 10.1016/j.bandc.2005.05.001. Epub 2005 Jun 21. PMID 15975700